CLINICAL TRIAL: NCT02903472
Title: Gastrointestinal (GI) and Urinary Tract (UT) Microbiome (MICRO) After Spinal Cord Injury (SCI)
Brief Title: Gastrointestinal and Urinary Tract Microbiome After SCI
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Praxis Spinal Cord Institute (Other)
Responsible Party: Principal Investigator, Matthias Walter, Principal Investigator, University of British Columbia
Other Study IDs: H16-00954
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Spinal Cord Injury
Keywords: SCI; microbiome; metabolome; GI; UTI; DNA; genomics; infections; tetraplegic; paraplegic
MeSH Terms: conditions — Spinal Cord Injuries; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and urine samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Acute to first year after SCI: Individuals sustained SCI within a 1-year period
- Chronic: Individuals sustained SCI more than1 year ago

SUMMARY:
Changes in the GI microbiota and/or metabolomics have been linked to evolving transformations in immune system function and infection rates in experimental SCI in animal models. A recent study involving chronic survivors of SCI show distinct GI microbiome changes in comparison to healthy controls. GI microbial metabolism of dietary components has been causally linked to various health conditions, such as cardiovascular disease, infections, which is an ongoing concern for chronic SCI survivors. It is probable that alterations of GI microbiota are established acutely after SCI and could subsequently alter medical care and impact health outcomes for people living with SCI.

This project is a pilot study to describe any changes in the GI and urinary tract microbiota as they appear over the first year after SCI. When available, data on factors, other than SCI, that may impact change in the gut microbiome after SCI will also be noted, including:

* the level and severity of SCI,
* the time since SCI,
* the person's immune profile,
* the antibiotic regimen of the individual and time since antibiotic administration,
* the incidence and type of infections after SCI and
* the person's diet or activities after SCI

DETAILED DESCRIPTION:
Study 1 - Acute to first year after SCI:

The investigators wish to recruit 4 types of SCI participants (~8 tetraplegic motor complete SCI participants, ~8 tetraplegic motor incomplete SCI, ~8 paraplegic motor complete SCI and ~8 paraplegic motor incomplete SCI). This totals 32 participants.

The investigators will non-invasively collect small (<1 gram) stool and urine (<1 ml) samples from people who have suffered an acute SCI and have been admitted to their hospital for care and treatment of their injury.

The investigators will track changes in the microbiota, microbiome and metabolome within the gastrointestinal (GI) tract of people after acute spinal cord injury (SCI) through the non-invasive collection of a small stool sample during normal bowel routines at baseline (within the first week after SCI). Subsequent samples would be obtained in the same non-invasive nature at approximately 1, 3, 6, and 12 months after SCI, as part of any daily (in-patient or at home, outpatient) bowel routine. The stool samples will be processed for genomic analysis to identify GI bacterial species and any changes in an individual's GI microbiota and/or dysbiosis during the first year after SCI. As SCI increases the incidence and prevalence of urinary tract infections (UTIs), the investigators will track alteration within the microbiota of the urinary tract to ascertain whether there are links in the bacterial taxa between the GI system and urinary tract.

------------------------------------------------------------------------------

Study 2 - Chronic:

This study will attempt to recruit ~ 20 chronic SCI participants with or without recurrent infections (e.g. UTI, skin or systemic) to ascertain whether there is a correlation between a dysbiotic microbiota presentation and recurrent infections.

A small stool or urine sample will be obtained at home by participants and subsequently collected for genomic analysis during a person's routine outpatient clinic visit.

All replicate data (3 samples per individual at 3 different time points - 1, 6 and 12 months post baseline visit) from chronic participants would be matched as much as possible for age, gender, diet, type of SCI, time since SCI, activity, and should only differ in terms of recurrent infections and antibiotic prescriptions. The goal here would be to characterize any gut microbiota differences between the two disparate groups. The data may guide the development of future studies to investigate treatment options. During chronic SCI, many recurrent infections are UTIs; thus, the investigators will also monitor differences between the two group in the microbiota and metabolomics of the urinary tract.

ELIGIBILITY:
INCLUSION CRITERIA ------------------------------------

* Participants with acute SCI

  * Male or Female of the age of majority in his or her province/state/country OR Minor between 16 y.o. and the age of majority with informed consent provided by participant and parent or guardian.
  * Tetraplegic or paraplegic motor complete SCI (AIS A, B) or motor incomplete SCI (AIS C, D) involving a single non-penetrating traumatic injury to the C2-S1 spinal cord, treated surgically or non-surgically.
  * Preferably participants will be admitted to a study center within 48 hours of SCI. However, participants can be included within 7 days post injury.
  * Able to provide informed consent.
  * Able to converse in the language native to the country where the hospital is located.
  * Have the capacity to follow the study procedure.
* Participants with chronic SCI

  * Male or Female of the age of majority in his or her province/state/country OR Minor between 16 y.o. and the age of majority with informed consent provided by participant and parent or guardian
  * Tetraplegic or paraplegic motor complete SCI (AIS A, B) or motor incomplete SCI (AIS C, D) involving a single non-penetrating traumatic injury to the C2-S1 spinal cord, treated surgically or non-surgically
  * Able to provide informed consent
  * Able to converse in the language native to the country where the hospital is located
  * Have the capacity to follow the study procedure

EXCLUSION CRITERIA ------------------------------------

* Participants with acute SCI

  * Spinal cord injury with sensory deficit only (i.e. no motor deficit)
  * Penetrating spinal cord injury (including gunshot wounds)
  * Associated head injury or other major cognitive deficit (i.e. condition where comprehension may be impaired such that informed consent process or outcome assessment cannot be completed with confidence)
  * Concomitant medical conditions associated with SCI that would interfere with informed consent process or outcome assessment
  * Pre-existing history of a chronic bowel disorder (e.g. Crohn's disease, ulcerative colitis)
  * Pre-existing history of:

    * recurrent infectious diseases (3 or more times a year), e.g. urinary tract infections, pneumonia
    * Immune disorders (e.g. rheumatoid arthritis, systemic lupus) or
    * neurodegenerative syndromes
  * Presence of a systemic disease that might interfere with the safety, compliance or assessments being used in this project (e.g., clinically significant cardiac disease, including chronic hypertension, HIV)
  * Any other medical condition that in the investigator's opinion would render the protocol procedures dangerous or impair the ability of the patient to participate in the study
  * Female participants who are pregnant
* Participants with chronic SCI

  * Spinal cord injury with sensory deficit only (i.e. no motor deficit)
  * Penetrating spinal cord injury (including gunshot wounds)
  * Associated head injury or other major cognitive deficit (i.e. condition where comprehension may be impaired such that informed consent process or outcome assessment cannot be completed with confidence)
  * Concomitant medical conditions associated with SCI that would interfere with informed consent process or outcome assessment
  * Pre-existing history of a chronic bowel disorder (e.g. Crohn's disease, ulcerative colitis)
  * Presence of a systemic disease that might interfere with the safety, compliance or assessments being used in this project (e.g., clinically significant cardiac disease, including chronic hypertension, HIV)
  * Any other medical condition that in the investigator's opinion would render the protocol procedures dangerous or impair the ability of the patient to participate in the study
  * Female participants who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from both the acute and chronic populations of people living with SCI, specifically those treated as either inpatients and/or outpatients.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in GI microbiota | one year
  Establishing the correlations between changes in neurological and functional capabilities in individuals with SCI and difference in the gut intestinal (GI) microbiota or metabolome and determining how such changes contribute to increased rates of infections

CONTACTS AND LOCATIONS:
Overall Officials: John Steeves, PhD, Principal Investigator — University of British Columbia; Matthias Walter, MD, PhD, Principal Investigator — University of British Columbia; Brett Finlay, PhD, Principal Investigator — University of British Columbia
Locations (6):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States
- Canada (2):
  - University of Calgary Department of Clinical Neurosciences, Calgary, Alberta
  - Stan Cassidy Center for Rehabilitation, Fredericton, New Brunswick
- Spinal Cord Injury Unit, Institut Guttmann Barcelona, Barcelona, Spain
- Balgrist University Hospital, Zurich, Switzerland
- Gaziler PMR, Training and Research Hospital, Department of PMR, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No